CLINICAL TRIAL: NCT07343544
Title: Estudio clínico Para Evaluar Los Efectos y la Seguridad de un Producto cosmético en Sujetos Con Signos de Envejecimiento cutáneo.
Brief Title: Clinical Trial to Assess the Efficacy and Safety of a Cosmetic Product in Individuals Showing Signs of Cutaneous Aging.
Acronym: SkinMeter
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Collaborators: Dr. Goya Análisis, SL. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB BIOTICS_2501_COS /SkinMeter
Record Dates: First submitted 2025-12-09; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Skin; Skin Ageing; Fine Lines; Face Aging/Photo Aging of Moderate Grade; Face Skin Photoaging
Keywords: Face Skin; Postbiotics; Skin; Skin ageing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Other): Open Label Active Product
  Interventions: Other: Active cream

INTERVENTIONS:
Other: Active cream — Active facial cream with postbiotics.

SUMMARY:
This clinical study investigates the effects and safety of a topical cosmetic product containing postbiotics (Bifida ferment extract and Pediococcus ferment extract) in women aged 35-60 with visible signs of skin aging.

The study is a 3-month, single-center, intra-subject controlled trial involving 45 Caucasian women with sensitive or normal skin. Participants will apply 1 ml of the product twice daily. Clinical evaluations will be conducted at baseline and at 1 month, 2 months, and 3 months, using validated dermatological scales and non-invasive instruments (AEVA3D, Mexameter®, MoistureMap®, Cutometer®, Tewameter®, Clarius®, Glossymeter®).

Safety will be assessed through systematic monitoring of adverse events, with serious adverse events expected to remain below 1%. Subjective perception will be evaluated via structured questionnaires.

DETAILED DESCRIPTION:
This clinical study is designed to evaluate the effects and safety of a topical cosmetic product formulated with postbiotic ingredients in adult women presenting visible signs of skin aging. The product contains Bifida ferment extract and Pediococcus ferment extract, selected for their scientifically supported properties in enhancing skin barrier function, reducing oxidative stress, and improving overall skin appearance.

The study is a prospective, single-center, intra-subject controlled clinical trial with a total duration of three months. Forty-five Caucasian women aged between 35 and 60 years will be enrolled. Participants must present mild to moderate facial wrinkles and/or pigmentation spots and will be evenly distributed between sensitive and normal skin types. Inclusion and exclusion criteria are clearly defined to ensure participant safety and data reliability.

Participants will apply 1 ml of the cosmetic product twice daily (morning and evening) to clean, dry facial skin. The study includes four scheduled visits: pre-selection, baseline (T0), (T1), 1 month (T2), 2 months (T3), and 3 months (T4). During these visits, clinical assessments will be conducted using validated dermatological scales (Skin Aging Atlas and Glogau scale) and non-invasive instrumental evaluations.

Instrumental assessments include AEVA3D, Mexameter®, MoistureMap®, Cutometer®, Tewameter®, Clarius®, Glossymeter®.

Photographic documentation will be performed using Visiofaceae, capturing standardized facial images at each visit.

Subjective perception will be evaluated through structured questionnaires administered at T1, T2, T3, and additionally at day 7. These questionnaires assess product appreciation, organoleptic characteristics, absorption, residue, and perceived effects on skin condition.

Safety monitoring includes systematic documentation of all adverse events (AEs). The expected incidence of SAEs related to the product is below 1%. All safety data will be recorded in the Case Report Form (CRF) and analyzed according to Good Clinical Practice (GCP) guidelines. Participants will be compensated for travel and related expenses.

Statistical analysis will be conducted using RStudio software. The study is powered to detect significant changes in skin aging parameters, with a sample size of 45 participants calculated to achieve 80% statistical power. Analysis will include descriptive statistics, repeated measures ANOVA, and mixed model repeated measures (MMRM) to evaluate treatment effects over time.

This study aims to provide robust clinical evidence supporting the efficacy and safety of a novel cosmetic formulation based on postbiotic technology, contributing to the development of innovative anti-aging skincare solutions.

ELIGIBILITY:
Inclusion Criteria:

* Female participants.
* Age between 35 and 60 years.
* All skin types (combination, oily, dry, and/or normal).
* Skin condition: 50% sensitive skin and 50% normal skin.
* Visible signs of facial skin aging (mild/moderate wrinkles and/or pigmentation spots).
* Willingness to participate voluntarily and provide written informed consent.
* Ability to understand the study objectives and procedures.
* Good general health (physical and mental).
* Availability to attend all scheduled visits at the research center.
* Discontinuation of anti-aging products on the experimental area (face) at least 7 days prior to study start.
* Commitment not to change facial hygiene routines during the study.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* History of allergy to cosmetic products and/or dietary supplements.
* Known allergy or hypersensitivity to any component of the product.
* History or current diagnosis of cancer.
* Active skin diseases or infections in the experimental area.
* Recent or planned surgical or aesthetic interventions in the experimental area Medical-aesthetic treatments on the face within the last 6 months (e.g., botulinum toxin, hyaluronic acid, laser, radiofrequency, HIFU, deep chemical peels, microneedling with actives).
* Relevant dermatological conditions in the experimental area (eczema, psoriasis, allergic/contact dermatitis, etc.).
* Use of topical or systemic medications affecting the skin (retinoids, antibiotics, corticosteroids) within the last 3 months.
* Current or planned use of supplements that may affect skin health (collagen, antioxidant vitamins A/C/E, zinc, omega-3, oral probiotics/prebiotics).
* Systemic diseases such as autoimmune disorders (rheumatoid arthritis, lupus, multiple sclerosis), chronic viral infections (HIV, hepatitis B/C), or severe metabolic diseases.
* Use of any product other than the study product on the experimental area during the study.
* Planned significant changes in health habits during the study (diet, physical activity, structured exercise programs).
* Recent or planned changes in hormonal contraceptives.
* Sun or UVA exposure during the study.
* Participation in another clinical study involving the same experimental area
* Application of any product on the experimental area on the day of study initiation.
* Any medical condition, at the investigator's discretion, that may interfere with protocol adherence or participant safety.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Wrinkle Reduction | From baseline to the end of treatment at 3 months
  Changes in visible signs of skin aging (wrinkles and spots) after 3 months of continuous application. Assess the evolution of wrinkles using AEVA3D-HE2.

SECONDARY OUTCOMES:
Spot Depigmentation | From baseline until the end of treatment at 3 months
  Evaluate the improvement in facial pigmentation using a clinical scale adapted from the Glogau Scale.
Facial Contour Evolution | From baseline until the end of treatment at 3 months
  Assess the evolution of contour after 1, 2, and 3 months using AEVA3D-HE2.
Spot Evolution | From baseline until the end of treatment at 3 months
  Assess the evolution of facial spots after 1, 2, and 3 months using Mexameter® MX 18.
Skin Hydration | From baseline until the end of treatment at 3 months
  Determine facial hydration after 1, 2, and 3 months using MoistureMap® MM200.
Firmness & Elasticity | From baseline until the end of treatment at 3 months
  Determine facial firmness and elasticity after 1, 2, and 3 months using Cutometer® MPA 580.
Barrier Function | From baseline until the end of treatment at 3 months
  Determine facial barrier function after 1, 2, and 3 months using Tewameter® TM 300.
Dermal Thickness | From baseline until the end of treatment at 3 months
  Changes in dermal thickness using Clarius® ultrasound.
Skin Radiance | From baseline until the end of treatment at 3 months
  Changes in facial radiance using Skin-Glossymeter® GL200.
Self-perceived improvement | From baseline until the end of treatment at 3 months
  Changes in self-perceived improvement assessed with subjective question.

CONTACTS AND LOCATIONS:
Overall Officials: Ester Moreno Artero, PhD, Principal Investigator — Dr. Goya Análisis

IPD SHARING:
Plan to Share IPD: No
Sponsor will evaluated IPD sharing upon request